CLINICAL TRIAL: NCT05795530
Title: Genetic Background of Hearing Loss and Vestibular Function Evaluation Following Cochlear Implantation
Brief Title: Vestibular Function in Cochlear Implants
Status: Completed | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Marketa Bonaventurova, Principle Investigator, Charles University, Czech Republic
Other Study IDs: CharlesUCZ
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Cochlear Trauma; Vestibular Disorder; Deafness, Bilateral
Keywords: cochlear implant
MeSH Terms: conditions — Vestibular Diseases; Hearing Loss, Bilateral | interventions — Cochlear Implantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cochlear implant recipients: 57 consecutive cochlear implant recipients
  Interventions: Procedure: cochlear implantation

INTERVENTIONS:
Procedure: cochlear implantation — surgery for bilateral hearing loss

SUMMARY:
The objective of this study is to identify possible preoperative risk factors including genetic background and to suggest the optimal test battery of vestibular function in cochlear implant recipients

DETAILED DESCRIPTION:
The objective of this study is to identify possible preoperative risk factors including genetic background and to suggest the optimal test battery of vestibular function in cochlear implant recipients Participants underwent standard vestibular testing including video head impulse test (vHIT), vestibular evoked myogenic potentials (VEMP), subjective visual vertical and stabilometry before and after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* profound bilateral sensorineural hearing loss meeting criteria for cochlear implantation

Exclusion Criteria:

* profound unilateral sensorineural hearing loss meeting criteria for cochlear implantation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 57 adult CI recipients The indication for surgery was hearing impairment. Round window approach was used preferably for insertion of the electrode array. Anamestic data as a history of hearing impairment, family history and the use of hearing aids were collected from all the patients.
  They underwent routine vestibular testing before and after the intervention.
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
vestibular function | from 2 days before the intervention to 3 weeks after the intervention
  semicircular canal function measured by vHIT
vestibular function | from 2 days before the intervention to 3 weeks after the intervention
  otolith function measured by VEMP
postural function | from 2 days before the intervention to 3 weeks after the intervention
  postural function and stability measured by stabilometry

CONTACTS AND LOCATIONS:
Overall Officials: Zuzana Balatkova, Study Chair — Dept Of ENT, 1st Faculty Of Medicine, University Hospital Motol
Locations (1):
- Department of Otorhinolaryngology and Head and Neck Surgery, 1st Faculty of Medicine Charles University and Motol University Hospital, Postgraduate Medical School, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No